CLINICAL TRIAL: NCT05857644
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO COMPARE THE PHARMACOKINETICS OF PF-07923568 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: A Study to Compare How the Study Medicine (PF-07923568) is Processed in Participants With Different Levels of Loss of Liver Function to Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5241012; NCT05857644 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-04-06; First posted 2023-05-12 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Liver Diseases; Hepatic Impairment
Keywords: healthy volunteers
MeSH Terms: conditions — Liver Diseases | interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: An open-label, single dose, parallel group, multicenter study to investigate the effect of varying degrees of hepatic function on the plasma PK of PF-07923568 after a single, oral 200 mg dose administered in the fed state (standard breakfast).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy subjects (Experimental): One time dose of 4 capsules taken orally.
  Interventions: Drug: PF-07923568
- Mild Hepatic impaired subjects (Experimental): One time dose of 4 capsules taken orally.
  Interventions: Drug: PF-07923568
- Moderate hepatic impaired subjects (Experimental): One time dose of 4 capsules taken orally
  Interventions: Drug: PF-07923568
- Severe Hepatic Impaired Subjects (Experimental): One time dose of 4 capsules taken orally.
  Interventions: Drug: PF-07923568

INTERVENTIONS:
Drug: PF-07923568 — One time dose of 4 capsules taken orally.
  Other Names: Sisunatovir

SUMMARY:
The purpose of this study is to learn how the study medicine (PF-07923568) is processed in participants with liver function loss compared to healthy participants. The different levels of liver function loss can be mild, moderate or severe.

This study is seeking participants who:

* are male or female of 18 years of age or older.
* are examined to be healthy (group with no loss of liver function).
* have mild, moderate, and severe liver disease (group with loss of liver function).

All participants will receive a one-time dose of 4 capsules of PF-07923568 which will be taken by mouth. All participants will remain at the study clinic for 6 days for safety review and laboratory collections. This is to see how the study medicine is being broken down by the liver over time.

All participants selected in the study will be required to go through a screening period up to 28 days. A screening period is the time during which a few participants are examined to see whether they are fit for the study. During this period, the participant's medical history and past and current medications will be reviewed. A series of tests will also be performed to see if they are good to be selected for the study. If the participant meets all required criteria and are interested in continuing, the participant will be brought into the study clinic to stay overnight for 6 days. On day 6, the participant will be discharged. About 28 to 35 days after discharge, the participant will be contacted for a follow up visit either in person or by telephone. This is to check up on how the participant is doing and to conclude the study.

ELIGIBILITY:
Inclusion Criteria: for healthy volunteers:

* BMI of 17.5 to 38.0 kg/m2, inclusive, and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.
* At screening, no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, including BP and pulse rate measurement, standard 12-lead ECG and clinical laboratory tests.
* body weight within +/-15 kg of the average of pooled hepatic impaired group and +/- 10 years of the average pooled hepatic impairment group.

  --Exclusion criteria for all participants:
* Any condition or surgery possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection)
* Positive HIV antibodies
* Positive drug or alcohol test eGFR <60 mL/min/1.73m2 at screening

Exclusion criteria for non-healthy participants who have hepatic impairment:

* Stable concomitant meds and hepatic impairment with no change in the last 28 days
* Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy (defined as <1 year).
* A diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, PE, liver biopsy, hepatic ultrasound, CT scan, or MRI.
* History of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 4 weeks prior to screening.

  --Severe ascites and/or pleural effusion, except for those categorized as severe hepatic impairment who may be enrolled provided participant is medically stable, per the investigators' medical judgment.
* Previously received a kidney, liver, or heart transplant. ALT/AST greater than 5X upper limit normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with varying degrees of hepatic function were enrolled in 4 groups
Groups:
- No Hepatic Impairment; Mild Hepatic Impairment; Moderate Hepatic Impairment; Severe Hepatic Impairment: Participants received an oral single dose of sisunatovir 200 mg (4 × 50 mg capsules) with the morning meal.
Period: Overall Study
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started (28) | 8 | 8 | 8 | 4
Completed (28) | 8 | 8 | 8 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 28
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 0 | 1 | 1 | 0 | 2
  45-64 years | 7 | 3 | 6 | 2 | 18
  ≥65 years | 1 | 4 | 1 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 1 | 12
  Male | 4 | 5 | 4 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 3 | 10
  Not Hispanic or Latino | 7 | 5 | 5 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Plasma Maximum Concentration (Cmax) of Sisunatovir Following Administration of a Single Oral Dose
Description: Cmax was the highest concentration observed directly from data
Time Frame: Hours 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, and 120 postdose from Day 1 to Day 6
Population: All participants who received at least 1 dose of sisunatovir and had at least 1 of the pharmacokenetic parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
Nanograms/milliliter (ng/mL) | 81.25 (57) | 68.52 (73) | 73.85 (73) | 127.8 (38)
Statistical Analysis 1: Comparison: No Hepatic Impairment vs Mild Hepatic Impairment; Test type: Other; Geometric mean ratio = 84.33, 90% CI 2-sided [50.94 to 139.59] — Mild Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 2: Comparison: No Hepatic Impairment vs Moderate Hepatic Impairment; Test type: Other; Geometric mean ratio = 90.89, 90% CI 2-sided [54.91 to 150.45] — Moderate Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 3: Comparison: No Hepatic Impairment vs Severe Hepatic Impairment; Test type: Other; Geometric mean ratio = 157.23, 90% CI 2-sided [84.81 to 291.49] — Severe Hepatic Impairment versus No Hepatic Impairment

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Sisunatovir Following Administration of a Single Oral Dose
Description: AUClast was determined using linear/Log trapezoidal method
Time Frame: Hours 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, and 120 postdose from Day 1 to Day 6
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
nanograms*hour/milliliter (ng*hr/mL) | 891.6 (37) | 732.6 (70) | 1166 (99) | 3437 (20)
Statistical Analysis 1: Comparison: No Hepatic Impairment vs Mild Hepatic Impairment; Test type: Other; Geometric mean ratio = 82.17, 90% CI 2-sided [49.24 to 137.11] — Mild Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 2: Comparison: No Hepatic Impairment vs Moderate Hepatic Impairment; Test type: Other; Geometric mean ratio = 130.82, 90% CI 2-sided [78.40 to 218.30] — Moderate Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 3: Comparison: No Hepatic Impairment vs Severe Hepatic Impairment; Test type: Other; Geometric mean ratio = 385.52, 90% CI 2-sided [205.92 to 721.77] — Severe Hepatic Impairment versus No Hepatic Impairment

3. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Sisunatovir Following Administration of a Single Oral Dose
Description: AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel was the terminalphase rate constant.
Time Frame: Hours 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, and 120 postdose from Day 1 to Day 6
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng*hr/mL | 922.6 (35) | 765.6 (68) | 1213 (95) | 3617 (19)
Statistical Analysis 1: Comparison: No Hepatic Impairment vs Mild Hepatic Impairment; Test type: Other; Geometric mean ratio = 82.99, 90% CI 2-sided [50.53 to 136.28] — Mild Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 2: Comparison: No Hepatic Impairment vs Moderate Hepatic Impairment; Test type: Other; Geometric mean ratio = 131.52, 90% CI 2-sided [80.09 to 215.99] — Moderate Hepatic Impairment versus No Hepatic Impairment
Statistical Analysis 3: Comparison: No Hepatic Impairment vs Severe Hepatic Impairment; Test type: Other; Geometric mean ratio = 392.10, 90% CI 2-sided [213.57 to 719.85] — Severe Hepatic Impairment versus No Hepatic Impairment

4. Secondary Outcome: Number of Participants With All-causality Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, Treatment-related TEAEs, and Discontinuations From Study Due to TEAEs
Description: Adverse event (AE) was any untoward medical occurrence in the participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Serious AE was any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or was considered to be an important medical event. Any events occurring following start of treatment or increasing in severity were counted as treatment-emergent. AEs included both serious and non-serious AEs.
Time Frame: Day -1 through follow-up (Day 29-36)
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
Participants
  All-causality TEAEs | 1 | 0 | 1 | 1
  Serious TEAEs | 0 | 0 | 0 | 0
  Treatment-related TEAEs | 1 | 0 | 1 | 0
  Discontinuations from study due to TEAEs | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, absolute and percent total neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen/urea and creatinine, fasting glucose, calcium, sodium, potassium, chloride, total carbon dioxide, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin and total protein), urinalysis (pH, qualitative glucose, qualitative protein, qualitative blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy, urinary albumin to creatinine ratio and urinary protein to creatinine ratio) and other tests. Abnormality was determined by the investigator. Only lab abnormalities with at least 1 occurrence in participants are reported.
Time Frame: Day -1 and Day 6
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention, and who had at least one observation of the given laboratory test and had a laboratory abnormality meeting specified criteria while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
Participants
  Erythrocytes <0.8 x lower limit of normal (LLN): number analyzed (Participants) | 8 | 7 | 8 | 4
  Erythrocytes <0.8 x lower limit of normal (LLN) | 0 | 0 | 0 | 2
  Ery. Mean Corpuscular Volume >1.1 x upper limit of normal (ULN): number analyzed (Participants) | 8 | 7 | 8 | 4
  Ery. Mean Corpuscular Volume >1.1 x upper limit of normal (ULN) | 0 | 0 | 0 | 2
  Ery. Mean Corpuscular Hemoglobin Concentration <0.9 x LLN: number analyzed (Participants) | 8 | 7 | 8 | 4
  Ery. Mean Corpuscular Hemoglobin Concentration <0.9 x LLN | 0 | 0 | 2 | 1
  Platelets <0.5 x LLN: number analyzed (Participants) | 8 | 7 | 8 | 3
  Platelets <0.5 x LLN | 0 | 0 | 0 | 1
  Lymphocytes <0.8 x LLN: number analyzed (Participants) | 8 | 7 | 8 | 4
  Lymphocytes <0.8 x LLN | 0 | 0 | 0 | 1
  Neutrophils < 0.8 x LLN: number analyzed (Participants) | 8 | 7 | 8 | 4
  Neutrophils < 0.8 x LLN | 0 | 0 | 0 | 1
  Activated Partial Thromboplastin Time >1.1 x ULN | 3 | 1 | 5 | 1
  Prothrombin Time >1.1 x ULN | 1 | 1 | 1 | 4
  Prothrombin Intl. Normalized Ratio >1.1 x ULN | 1 | 0 | 1 | 3
  Bilirubin >1.5 x ULN | 0 | 0 | 0 | 3
  Direct Bilirubin > 1.5 x ULN: number analyzed (Participants) | 0 | 4 | 5 | 3
  Direct Bilirubin > 1.5 x ULN | 0 | 0 | 0 | 2
  Indirect Bilirubin >1.5 x ULN: number analyzed (Participants) | 0 | 4 | 5 | 3
  Indirect Bilirubin >1.5 x ULN | 0 | 0 | 0 | 2
  Gamma Glutamyl Transferase >3.0 x ULN | 0 | 0 | 3 | 0
  Albumin <0.8 x LLN | 0 | 0 | 0 | 2
  Potassium <0.9 x LLN | 0 | 0 | 0 | 1
  Bicarbonate <0.9 x LLN | 0 | 0 | 0 | 1
  Glucose - FASTING >1.5 x ULN | 0 | 0 | 1 | 0
  pH >8: number analyzed (Participants) | 8 | 8 | 7 | 4
  pH >8 | 0 | 0 | 1 | 1
  URINE Glucose ≥1: number analyzed (Participants) | 8 | 8 | 7 | 4
  URINE Glucose ≥1 | 0 | 0 | 1 | 0
  Urobilinogen ≥1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Urobilinogen ≥1 | 0 | 0 | 0 | 1
  Nitrite ≥1: number analyzed (Participants) | 8 | 8 | 7 | 4
  Nitrite ≥1 | 0 | 0 | 1 | 1

6. Secondary Outcome: Number of Participants With Vital Signs Meeting Categorical Criteria
Description: Supine blood pressure and pulse rate were measured. Categorical classes for vital signs of potential clinical concerns were defined as followed: systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); diastolic blood pressure (DBP) <50 mmHg; pulse rate <40 beats per minute (bpm); pulse rate >120 bpm, and increase from baseline in SBP ≥30 mmHg; decrease from baseline in SBP ≥30 mmHg; increase from baseline in DBP ≥20 mmHg; decrease from baseline in DBP ≥20 mmHg. The baseline measurement was the predose measurement on Day 1. Changes from baseline was defined as the change between the postdose and baseline measurements.
Time Frame: Day -1, Day 1, Day 2, and Day 6
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
Participants
  DBP: increase from baseline ≥20 mmHg | 0 | 1 | 0 | 0
  DBP: decrease from baseline ≥20 mmHg | 0 | 0 | 1 | 0
  SBP <90 mmHg | 1 | 0 | 1 | 0
  SBP: increase from baseline ≥30 mmHg | 0 | 1 | 1 | 0

7. Secondary Outcome: Number of Participants With Electrocardiograms (ECGs) Meeting Categorical Criteria
Description: Number of participants with ECG findings meeting the following criteria: time between the onset of atrial depolarization and onset of ventricular depolarization (PR interval) ≥300 msec; time from ECG Q-wave to the end of the S wave corresponding to ventricular depolarization (QRS duration) ≥140 msec; correct time from ECG Q-wave to the end of the T wave corresponding to electrical systole for heart rate using Fridericia's formula (QTcF interval): ≥450 to <480 msec; QTcF interval ≥480 to <500 msec; QTcF interval: ≥500 msec; PR interval percent change from baseline (≥25/50%): ≥25% if baseline >200 msec or ≥ 50% if baseline ≤200 msec; QRS duration percent change from baseline ≥50%; QTcF interval change from baseline: >30 to ≤60 msec; QTcF interval change from baseline >60 msec. The baseline measurement was the predose measurement on Day 1. Changes from baseline was defined as the change between the postdose and baseline measurements.
Time Frame: Day -1, Day 1, Day 2, and Day 6
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
Participants
  QTcF interval: ≥450 msec to <480 msec | 0 | 1 | 1 | 3
  QTcF interval: ≥480 msec to <500 msec | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day -1 through follow-up (Day 29-36)
Description: The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant beginned from the time the participant provides informed consent, which was obtained before before undergoing any study-related procedure and/or receiving study intervention, through and including a minimum of 28 calendar days, after the last administration of the investigational product.
Arm/Group | No Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 1/8 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Hepatic Impairment (N=8) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Severe Hepatic Impairment (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT05857644/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05857644/SAP_001.pdf